CLINICAL TRIAL: NCT03912649
Title: A Prospective, Single-centre, Non-comparative Feasibility Investigation to Evaluate Performance and Safety of RemovAid ™ Retrieval Device When Used for Removal of Palpable Subdermal Contraceptive Rod Implants
Brief Title: Investigation to Evaluate Performance and Safety of RemovAid ™ in Removal of Contraceptive Implants
Acronym: REVALID03
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Although the defined success rate needed for continuation of the investigation was met, due to the overall low success rate; it was considered, particularly considering the ongoing pandemic, to discontinue the investigation prematurely.
Sponsor: RemovAid AS (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REVALID03
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Removal Contraceptive Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RemovAid arm (Experimental): RemovAid arm -
  All subjects have their implant removed by the RemovAid device
  Interventions: Device: RemovAid

INTERVENTIONS:
Device: RemovAid — The RemovAid device is used for removal

SUMMARY:
The safety and efficacy of a subdermal implant retrieval device (RemovAid) is investigated in a population of 25 women seeking removal of their palpable contraceptive implants.

The primary endpoint of the device is to evaluate the performance of the device, specifically its success rate in removing palpable contraceptive implants. The device shall be able to fixate at least 80% of palpable implants, and successfully remove at least 90% of these implants.

DETAILED DESCRIPTION:
Similar to the REVALID and REVALID02 investigations, the REVALID03 investigation aims to recruit a total of 25 women with a palpable contraceptive implant due for removal, in order to obtain at least 20 successful fixations.

The implant retrieval device aims to standardize and simplify the implant removal procedure. There is no comparator in the investigation. Descriptive data will be recorded, all recruited subjects will be exposed to the investigational medical device (IMD) The primary endpoint is the percentage of fixated implants that are successfully removed without the use of additional tools.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Willing to remove a palpable subdermal Implanon/ Nexplanon CI
* Willing and able to give written informed consent for participation in the investigation
* Willing to provide follow-up information according to the Clinical Investigators brochure

Exclusion Criteria:

* Known allergy to local anaesthetic (lidocaine/lignocaine) or disinfectant (chlorhexidine).
* Active skin lesion over the CI.
* The Investigator considers the subject unlikely to comply with investigational procedures, restrictions and requirements.
* Any contraindication for removal of the PI, as judged by the Investigator.
* Any disorders or medications that might affect coagulation, as judged by the Investigator.
* Any conditions suspected to affect healing or increase risk of infection (e.g. keloid tendency, diabetes or any upper arm dermatological condition that may affect upper arm healing)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Successful removal of implant | 15 minutes
  The percentage of fixated implants that are successfully removed by the device without the use of additional tools

SECONDARY OUTCOMES:
Frequency, severity, causality and outcome of adverse events (AEs) | 1 week
  Both Anticipated and unanticipated AEs will be recorded, both immediately following the intervention and at follow-up
Pain during procedure: Visual Analogue Scale | 15 minutes
  Mean pain score (maximum pain intensity during the procedure) indicated by the subject on a Visual Analogue Scale 0-100 mm ruler, assuming that anaesthesia has been properly administered. Higher values represent a worse outcome.
Success of fixation of implant | 5 minutes
  Percentage of palpable implants where the implant could be seen and/or felt on both sides of the clamp after maximum three attempts of fixation. 80% or more is considered success.
Duration of procedure | 25 minutes
  Mean time from making incision until implant is removed, and first touching subject with the device until implant extracted
Technical functionality of device determined by an operators questionnaire | 5 minutes
  Fulfilment of pre-defined technical requirements, as documented on an operator functionality questionnaire. The questionnaire consists of a range of yes/no questions to device functionality
Operators impression of the device | 5 minutes
  The operator's global impression of the IMD will be assessed using a scale 1-5, where 5 is excellent and 1= poor
Subject satisfaction: 5- point scale | 5 minutes
  The subject's global assessment of satisfaction with the procedure will be assessed using a scale of 1-5, where 5 is excellent

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell-Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Adolescent Health Care Long-Acting Reversible Contraception Working Group, The American College of Obstetricians and Gynecologists. Committee opinion no. 539: adolescents and long-acting reversible contraception: implants and intrauterine devices. Obstet Gynecol. 2012 Oct;120(4):983-8. doi: 10.1097/AOG.0b013e3182723b7d. PMID 22996129
- [Background] Mansour D, Mommers E, Teede H, Sollie-Eriksen B, Graesslin O, Ahrendt HJ, Gemzell-Danielsson K. Clinician satisfaction and insertion characteristics of a new applicator to insert radiopaque Implanon: an open-label, noncontrolled, multicenter trial. Contraception. 2010 Sep;82(3):243-9. doi: 10.1016/j.contraception.2010.04.007. Epub 2010 May 18. PMID 20705152
- [Background] Mommers E, Blum GF, Gent TG, Peters KP, Sordal TS, Marintcheva-Petrova M. Nexplanon, a radiopaque etonogestrel implant in combination with a next-generation applicator: 3-year results of a noncomparative multicenter trial. Am J Obstet Gynecol. 2012 Nov;207(5):388.e1-6. doi: 10.1016/j.ajog.2012.08.002. Epub 2012 Aug 10. PMID 22939402
- [Background] Webb AM. Why go to Tiger Country? A report of two cases of Implanon removal. J Fam Plann Reprod Health Care. 2006 Jul;32(3):193-4. doi: 10.1783/147118906777888233. No abstract available. PMID 16857083
- [Background] Levine JP, Sinofsky FE, Christ MF; Implanon US Study Group. Assessment of Implanon insertion and removal. Contraception. 2008 Nov;78(5):409-17. doi: 10.1016/j.contraception.2008.06.016. Epub 2008 Sep 18. PMID 18929739
- [Background] Funk S, Miller MM, Mishell DR Jr, Archer DF, Poindexter A, Schmidt J, Zampaglione E; Implanon US Study Group. Safety and efficacy of Implanon, a single-rod implantable contraceptive containing etonogestrel. Contraception. 2005 May;71(5):319-26. doi: 10.1016/j.contraception.2004.11.007. PMID 15854630